CLINICAL TRIAL: NCT02025309
Title: Does Intraoperatively Administered Methylprednisolone Prolong the Neuromuscular Blocade Reversal Effect of Sugammadex?
Brief Title: Intraoperative Methylprednisolone and Sugammadex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Basak Ceyda MECO, MD, DESA, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 16-627-13
Record Dates: First submitted 2013-12-24; First posted 2014-01-01 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Neuromuscular Monitoring; Sugammadex Effect
Keywords: train of four; neuromuscular recovery; sugammadex
MeSH Terms: interventions — Neuromuscular Monitoring

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Methylprednisolone (Active Comparator): Patient in this group received general anaesthesia for surgical procedures. During the anesthesia management methylprednisolone was administered intravenously (1mg/kg) to the patients in this group. Also neuromuscular monitorisation was performed to assess the train of four ratio at the end of the procedure, after the reversal of neuromuscular block. All patients were followed during the recovery period from general anaesthesia and the time needed to regain a full neuromuscular recovery was noted. For that, the train of four ratio was followed up and the ratio of 0.9 was recorded.
  Interventions: Device: Neuromuscular monitorisation
- Group Control (Placebo Comparator): Patients who received general anaesthesia and endothracheal entubation but who did not recieved methyprednisone during general anaesthesia were enrolled in the study as control group. Neuromuscular monitorisation was performed to assess the train of four ratio at the end of the procedure, after the reversal of neuromuscular block. All patients were followed during the recovery period from general anaesthesia and the time needed to regain a full neuromuscular recovery was noted. For that, the train of four ratio was followed up and the ratio of 0.9 was recorded.
  Interventions: Device: Neuromuscular monitorisation

INTERVENTIONS:
Device: Neuromuscular monitorisation
  Other Names: Train of Four

SUMMARY:
Sugammadex, a modified γ-cyclodextrin is a selective relaxant-binding agent that reverses the effects of steroidal neuromuscular blocking agents, rocuronium and vecuronium. It shows its activity by encapsulating these. Likewise, some other steroid hormones and drugs like flucloxacillin, toremifene, fusidic acid can also be effected. Thus, assuming that methylprednisolone would also be encapsulated by sugammadex and decrease its efficiency, in this study we aimed to compare the recovery times from recuronium-induced muscle relaxation after reversal with sugammadex between patients who receive intraoperative methylprednisolone or not.

After institutional review board (IRB) approval and informed consent, 100 patients will be enrolled in this prospective, single center, controlled study. Anaesthesia will be induced with propofol (3mg/kg) and rocuronium (0.6 mg/kg), followed by sevoflurane maintenance. Patients will be divided randomly into two groups methylprednisolone administered group and control group respectively). Neuromuscular blockade will be monitored using calibrated acceleromyography train-of-four (TOF WATCH SX Organon Ltd, Dublin, Ireland). Once rocuronium-induced neuromuscular blockade recovers spontaneously to TOF-count-two, all patients will receive 2.0 mg/kg of sugammadex. Neuromuscular monitoring will be continued until recovery of the TOF ratio to 0.9 at the ulnar nerve. The time to recovery of TOF to 0.9 will be compared in both groups. The statistical analyses will be performed using Student T Test and Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* patient operated under general anesthesia and endothracheal intubation.
* 18-65 years old
* ASA II

Exclusion Criteria:

* Neuromuscular desease
* Renal desease
* Liver failure
* Hypersensitivity to the medications used in the study.
* Being on steroid medication
* Pregnanacy, Lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Train of four ratio 0.9 | During the procedure period.
  At the end of the procedure, train of four (TOF) monitorisation was continued and once rocuronium-induced neuromuscular blockade recovered spontaneously to TOF-count-two, all patients received 2.0 mg/kg of sugammadex. Then, neuromuscular monitoring was continued until recovery of the TOF ratio to 0.9 at the ulnar nerve. The time needed for the recovery of TOF to 0.9 was noted.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Hayriye Kocaoglu, MD, Principal Investigator — Ankara University Faculty of Medicine
Locations (1):
- Ankara University Faculty of Medicine, Ibni Sina Hospital OR, Ankara, Turkey (Türkiye)